CLINICAL TRIAL: NCT00518219
Title: To Compare the Efficacy and Safety of TW vs Valsartan in the MN
Brief Title: To Compare the Efficacy and Safety of Tripterygium Wilfordii (TW) Versus Valsartan in the Membranous Nephropathy (MN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0702
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-03

CONDITIONS: Membranous Nephropathy
Keywords: TW; Valsartan; treatment; membranous nephropathy; proteinuria
MeSH Terms: conditions — Glomerulonephritis, Membranous; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immunosuppressor (Experimental): TW 120mg/d，Valsartan,160mg/d
  Interventions: Drug: TW

INTERVENTIONS:
Drug: TW — TW,120mg/d
  Other Names: TW,Tripterygium wilfordii Hook.f

SUMMARY:
The purpose of this study is to assess the efficacy of TW compared to Valsartan in treatment of heavy proteinuria of membranous nephropathy.

DETAILED DESCRIPTION:
Membranous nephropathy with heavy proteinuria have high risks of progressing to CRF.

Tripterygium (TW) is a Chinese traditional patent drugs, it can reduce proteinuria of chronic glomerular nephritis,such as IgA nephropathy. So, we designed this randomized, prospective clinical trial to assess the efficacy and safety of TW versus Valsartan in the treatment of heavy proteinuria of MN.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven idiopathic membranous nephropathy
* Nephrotic syndrome with proteinuria (> 4 g/day) and serum albumin < 30 g/dl
* Age over 18 with informed consent

Exclusion Criteria:

* Patient with abnormal liver function tests
* Prior therapy with sirolimus, CSA, MMF, tacrolimus or azathioprin, chlorambucil, levamisole, methotrexate, or nitrogen mustard in the last 90 days,
* Active/serious infection,
* Patient with hepatitis B surface antigen or who is hepatitis C antibody positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To access the efficacy of TW compared to ARB in treatment of heavy proteinuria of membranous nephropathy | 12 months

SECONDARY OUTCOMES:
To investigate the safety and tolerability of TW vs ARB in treatment of MN | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Master, Principal Investigator — Jinling Hospital, China
Locations (1):
- Research Institute of Nephrology, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952